CLINICAL TRIAL: NCT05911815
Title: Evaluation Of The Diagnostic Role Of Hysterosalpingography In Cesarean Scar Niche Diagnosed By Hysteroscopy
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abdallah Saleh, Resident at gynecology department, Ain Shams University
Other Study IDs: AinG6/2023
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Radiation: hysterosalpingography — hysterosalpingogram (HSG) is an X-ray visualization of the lumen of the uterus and fallopian tubes, which can detect abnormalities including blockage, polyps, and salinities

SUMMARY:
The term CS niche (defect) describes the presence of a hypoechoic area within the myometrium in the isthmus (lower uterine segment) with discontinuation of myometrium at the site of previous CS. Hysterosalpingography is an important component in the diagnostic evaluation of the infertile woman. The number of hysterosalpingography examinations performed has significantly increased in recent years, likely due to the trend for women delaying pregnancy until later in life and the popularity of technical advances achieved in reproductive medicine.The term CS niche (defect) describes the presence of a hypoechoic area within the myometrium in the isthmus (lower uterine segment) with discontinuation of myometrium at the site of previous CS. The main purpose of the study is to evaluate the diagnostic role of HSG to early detect cesarean scar niche. To evaluate diagnostic role of hysterosalpingography (HSG) in cesarean scar niche at Early Cancer Detection and Gynecological Endoscopy Unit at Ain Shams Maternity Hospital within 6 months.

ELIGIBILITY:
Inclusion Criteria

* Age more than 18 years.
* Previous history of cesarean delivery.
* Cesarean scar niche confirmed by Hysteroscopy.
* Premenopausal status

Exclusion Criteria:

* Pregnancy.
* Contrast allergy.
* Active pelvic infection.
* Medical history interfering with HSG.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women undergoing Office Hysteroscopy at Early cancer Detection and Gynecological Endoscopy Unit at Ain Shams Maternity Hospital was checked to meet the inclusion criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Cesarean section niche appearance | baseline, pre-intervention
  The ability of hysterosalpingography to detect the cesarean section niche appearance

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams U, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No